CLINICAL TRIAL: NCT06391710
Title: A Multicenter, Randomized, Double-blind, Placebo-parallel-controlled, Phase II Clinical Study to Evaluate the Efficacy and Safety of HRS9531 Injection in Obese Subjects With Heart Failure With Preserved Ejection Fraction
Brief Title: HRS9531 Injection in Obese Subjects With Heart Failure With Preserved Ejection Fraction
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Shengdi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS9531-205
Record Dates: First submitted 2024-04-25; First posted 2024-04-30 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Heart Failure With Preserved Ejection Fraction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HRS9531 (Experimental)
  Interventions: Drug: HRS9531
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HRS9531 — subcutaneous
  Arms: HRS9531
Drug: Placebo — subcutaneous
  Arms: Placebo

SUMMARY:
This was a multicenter, randomized, double-blind, placebo-parallel-controlled Phase II clinical study to evaluate the efficacy and safety of HRS9531 Injection compared to placebo in obese subjects with heart failure with preserved ejection fraction.

A total of 200 obese subjects with heart failure with preserved ejection fraction would be enrolled. Eligible subjects were randomly assigned to either HRS9531 group or placebo group and were treated with HRS9531 injection or placebo, respectively, for 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age above or equal to 18 years at the time of signing informed consent.
2. Body mass index (BMI) greater than or equal to 28.0 kg/m^2
3. New York Heart Association (NYHA) Class II-IV;
4. Left ventricular ejection fraction (LVEF) greater than or equal to 45 percentage at screening

Exclusion Criteria:

1. Medical history of myocardial infarction, acute decompensated heart failure, heart failure requiring hospitalization or urgent heart failure visit, unstable angina, stroke, or transient ischemic attack within 30 days prior to or at screening;
2. Haemoglobin A1c (HbA1c) greater than or equal to 11.0% at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2024-05-06 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Change in KCCQ (Kansas City Cardiomyopathy Questionnaire) clinical summary score | From baseline (week 0) to week 36
Change in body weight | From baseline (week 0) to week 36

SECONDARY OUTCOMES:
Hierarchical composite of time to all-cause death | From baseline (week 0) to week 36,52
Hierarchical composite of number of heart failure events requiring hospitalisation or urgent heart failure visit | From baseline (week 0) to week 36,52
Hierarchical composite of time to the first heart failure events requiring hospitalisation or urgent heart failure visit | From baseline (week 0) to week 36,52
Hierarchical composite of difference at least 5 in KCCQ clinical summary score change from baseline to 36, 52 weeks | From baseline (week 0) to week 36,52
Change in KCCQ clinical summary score | From baseline (week 0) to week 52
Change in body weight | From baseline (week 0) to week 52
Change in C-Reactive Protein (CRP) | From baseline (week 0) to week 36,52
Change in N-terminal pro-b-type natriuretic peptide (NT-proBNP) | From baseline (week 0) to week 36,52

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided